CLINICAL TRIAL: NCT04821050
Title: A Randomized, Sham-Controlled, Double-Blind Study of Sacral Nerve Stimulation for Mild-to-Moderate or Refractory Rheumatoid Arthritis
Brief Title: Sacral Nerve Stimulation for Mild-to-Moderate or Refractory Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202002053
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Sacral nerve; Sacral nerve stimulation; Neuromodulation; randomized clinical trial; drug refractory
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Sacral nerve stimulation
  Interventions: Device: Sacral nerve stimulation
- Control (Sham Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Sacral nerve stimulation — A senior acupuncture doctor will pierce filiform needles through the sacral foramen into the S3 and S4 sacral nerves. These sites correspond to the Zhongliao and Xialiao acupoints in Traditional Chinese Medicine.
  Electrodes will be clamped on the filiform needles and an electrical current of 0.5 mA will be delivered. The stimulation will last for 60 minutes every time, once a day for 2 weeks.
  Arms: Treatment
Device: Sham stimulation — Shallow acupuncture stimulation will be performed at sites 8-10cm away from the acupoints in Group 1.
  Electrodes will be clamped on the filiform needles and an electrical current of 0.5 mA will be delivered. The stimulation will last for 60 minutes every time, once a day for 2 weeks.
  Arms: Control

SUMMARY:
This pilot study will assess the efficacy of sacral never stimulation (SNS) for the treatment of adult patients with active, mild-to-moderate rheumatoid arthritis or those with refractory disease. The study will enroll 60 subjects in a single center. All eligible subjects will be randomly divided into two groups at a ratio of 1:1. Half of the subjects will receive SNS (treatment) and the other half will receive sham stimulation (control). Subjects will be followed up for 2-4 weeks, according to their response to the treatment. Disease activity score, patient report outcomes and serum inflammatory cytokines will be observed before and after treatment.

DETAILED DESCRIPTION:
Studies have shown that vagus nerve stimulation (VNS) may exert an anti-inflammatory effect through mechanisms like cholinergic anti-inflammatory pathway (CAP). This anti-inflammatory function of VNS has been verified in collagen induced arthritis (CIA) rats, RA patients, and animal models of inflammatory bowel disease (IBD). In recent years, it was reported that sacral nerve stimulation (SNS) is a safer way to exert a similar anti-inflammatory effect as VNS. Therefore, this study aims to explore the therapeutic effect of SNS on RA patients.

This is a randomized controlled clinical trial which will enroll 60 eligible RA patients. These subjects will be divided into two groups at a ratio of 1:1, the treatment group (Group 1) who will receive SNS and the control group (Group 2) who will receive sham stimulation. The patients will lie in prone position. In Group 1, a senior acupuncture doctor will pierce filiform needles through the sacral foramen into the S3 and S4 sacral nerves. These sites correspond to the Zhongliao and Xialiao acupoints in Traditional Chinese Medicine. In Group 2, shallow acupuncture stimulation will be performed at sites 8-10cm away from the acupoints in Group 1. In both groups, electrodes will be clamped on the filiform needles and an electrical current of 0.5 mA will be delivered. The stimulation will last for 60 minutes every time, once a day for 2 weeks. If the subjects respond to the treatment well, SNS treatment will be continued for 2 weeks. The following parameters will be measured before and 2-4 weeks after treatment:

1. Disease activity-related indexes of RA: swelling joint number (SJC), tender joint number (TJC), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP);
2. Serum levels of inflammatory cytokines, including IL-6, IL-17, TNF-α, etc;
3. Patient report outcomes: Visual Analogue Scale (VAS) pain score, Health Assessment Questionnaire Disability Index (HAQ-DI) ;
4. Indexes of autonomic nervous function: serum level of norepinephrine (NE), heart rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age at screening
* Met the American College of Rheumatology criteria (2010) for RA
* Active mild to moderate RA (defined as 3.2 < DAS28-CRP< 5.1) naïve to any medication; or refractory RA who demonstrated an inadequate response or loss of response to 2 or more conventional synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) after treatment for at least 6 months.

Exclusion Criteria:

* Any severe chronic or uncontrolled comorbid disease, such as important organ failure, degree II and III heart block, clinically significant cardiovascular disease, severe infection, tumor, etc;
* Combined with other connective tissue diseases
* Cognitive impairment and can't cooperate
* Pregnancy or breastfeeding
* Bleeding or coagulation disorders
* Localized skin infections
* Intra-articular corticosteroid or pulse steroid within 2 weeks preceding the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The American College of Rheumatology (ACR) 20 response at Week 2 from Day 0 | Week 2
  Difference between treatment and control groups in the proportion of subjects who achieve at least 20% improvement from baseline to Week 2 in tender and swollen joint counts of 28 joints (scale 0=best to 28=worse) and 3 out of the following 5 measures: Health Assessment Questionnaire Disability Index (HAQ-DI) score (scale 0=no difficulty to 3=unable to do), subject global assessment (0=best to 10=worse), subject pain (0=no pain to 10=worse), evaluator's global assessment (0=best to 10=worse), or high sensitivity C-reactive protein (hsCRP) concentration (mg/mL) with higher values representing worse outcome.

SECONDARY OUTCOMES:
1. The Disease Activity Score 28-C-reactive protein (DAS28-CRP) good or moderate response as defined by European League Against Rheumatism (EULAR) | week 2
  The DAS28-CRP good or moderate response as defined by EULAR based on a composite score of 4 items: tender and swollen joint counts of 28 joints (scale 0=best to 28=worse), subject global assessment (0=best to 10=worse) and high-sensitivity C-reactive protein (hsCRP) concentration (mg/L) with higher values representing worse outcome
DAS28-CRP response (MCID -1.2) at Week 2 | wee 2
  DAS28-CRP response based on the minimal clinically important difference (MCID) of -1.2 from baseline
3. Health Assessment Questionnaire Disability Index (HAQ-DI) response (MCID -0.22) | week 2
  HAQ-DI response based on the MCID of -0.22 from baseline
Pain Visual Analogue Scale (scoring range 0 ~ 10) | week 2
  Changes from baseline to week 2.

CONTACTS AND LOCATIONS:
Overall Officials: Minning Shen, associate professor, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Dinglei Su, Nanjing, Jiangsu, China